CLINICAL TRIAL: NCT00237419
Title: An Open Label Extension, Investigator Initiated Trial to Examine Radiographic Progression , Efficacy and Safety of Long-Term Treatment With Infliximab in Patients With Ankylosing Spondylitis. EASIC (European Ankylosing Spondylitis Infliximab Cohort)
Brief Title: Examination of Radiographic Progression, Efficacy and Safety of Long-Term Treatment With Infliximab in Patients With Ankylosing Spondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rheumazentrum Ruhrgebiet (Other)
Collaborators: Centocor BV (Industry); Trial Coordination Center, 9713 GZ Groningen (Unknown); PPD Development, LP (Industry)
Responsible Party: Prof. Dr. Jürgen Braun, Rheumazentrum Ruhrgebiet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EASIC 30505
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Long-term therapy with infliximab; Radiographic progression
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

INTERVENTIONS:
Drug: infliximab — Infliximab infusions 5 mg/kg body-weight each 6 to 8 weeks

SUMMARY:
Ankylosing spondylitis (AS) is a chronic inflammatory disease that involves the sacroiliac joints, axial skeleton, entheses and peripheral joints. Current therapy for AS is mainly NSAIDs and physiotherapy which are oft insufficient. Treatment with the TNF-alpha blocking agent infliximab was shown to have definite clinical efficacy in patients with active AS on a short- and a long-term-basis over 2 years. We want to show that treatment with infliximab on a long-term basis over 4 years is safe and efficient and can prevent radiographic progression over a long period of time. Further we want to learn about the outcome after discontinuation of anti-TNF-alpha therapy.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic inflammatory disease of unknown etiology that involves the sacroiliac joints, axial skeleton, entheses and peripheral joints. Chronic inflammation of entheses leads to new bone formation, syndesmophytes and ankylosis of joints, primarily in the axial skeleton. This leads to a dramatic loss of range of motion and to disability. The disease may also have nonskeletal manifestations including uveitis, carditis, pulmonary fibrosis and cardiac conduction abnormalities.

Current therapy for AS is mainly with NSAIDs and physiotherapy which are often insufficient. Clinical outcome with conventional therapies has not been good, with 50-70% of patients progressing to fusion of the spine by 10 to 15 years. Treatment with the TNF-alpha blocking agent infliximab was shown to have definite clinical efficacy in patients with active ankylosing spondylitis on a short- and a long-term basis over 2 years.

There is limited data available on the efficacy and safety of long-term anti-TNF therapy for 3 and more years, the outcome after discontinuation of anti-TNF therapy and the effect of anti-TNF therapy on radiographic progression over a long period of time.

The ASSERT trial was a 2 year international randomized placebo controlled trial to evaluate the efficacy and safety ot treatment with infliximab in patients with active and severe AS. The EASIC trial is initiated to follow the European participants of the ASSERT trial for at least an additional 2 years of treatment combined with systematic data collection.

ELIGIBILITY:
Inclusion Criteria:

* All patients in Europe who have completed visit "week 96" of ASSERT (last infusion of infliximab)
* Capacity to understand and sign an informed consent form
* Capacity to read and understand subject assessment forms
* Using adequate birth control measures for the duration of the study and for 6 months after receiving the last infusion, if the patient is of childbearing potential
* Serum creatinine < 1,4 mg/dl
* Hemoglobin > 9,0 mg /dl for males and > 8,5 mg/dl for females
* Serum transaminase levels within 3 times the upper limit of normal range

Exclusion Criteria:

* Have used systemic prednisolone > 20 mg during the 2 weeks prior to screening
* Have used cytotoxic drugs after the end of ASSERT including chlorambucil, cyclophosphamide and alkylating agents
* Have received any previous treatment with etanercept or any other anti-TNF agent (other than infliximab) after the end of the ASSERT trial
* General medical exclusion criteria
* Use of any investigational drug within 30 days prio to screening
* Concomitant diagnosis or history of congestive heart failure
* History of latent or active tuberculosis
* Signs or symptoms suggestive of active tuberculosis
* Recent close contact with a person with active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2005-12; Primary Completion 2010-11 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Degree of structural damage (radiographic progression)after 4 and 6 years of infliximab therapy (2 years of ASSERT trial plus 2 years of EASIC trial) | November 2008 and November 2010

SECONDARY OUTCOMES:
Proportion of patients which have received anti-TNF-alpha therapy as standard care after the end of ASSERT | November 2005
Description of the various treatment regimens after the end of ASSERT of the participating AS patients in various countries | November 2005
Degree of spinal inflammation analyzed by MRI after discontinuation of infliximab and 4-8 weeks and 2 and 4 years after re-treatment | November 2010
Long-term efficacy of infliximab over 4 and 6 years of therapy measured by the ASAS response criteria | November 2010
Efficacy and safety of a new start of infliximab therapy after discontinuation for several months after 2 and 4 years of continuous treatment | November 2008 and November 2010
Long-term effects on QoL | November 2010
Long-term effects on health resource utilisation and productivity in paid and unpaid work | November 2010

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Braun, Prof. Dr., Principal Investigator — Rheumazentrum Ruhrgebiet
Locations (15):
- Belgium (4):
  - Erasme University Hospital, Brussels
  - Limburg University Centre, Diepenbeek
  - Universitair Ziekenhuis, Afdeling Rheumatologie, Ghent
  - University Hospital Leuven, Leuven
- University Central Hospital, Division of Rheumatology, Helsinki, Finland
- France (2):
  - Groupe Hopitalier Cochin, Paris
  - Universitat R. Descartes, Hopital Cochin, Paris
- Germany (4):
  - Charite Mitte, Berlin
  - Charite Klinikum Steglitz, Berlin
  - Rheumazentrum Ruhrgebiet, Herne
  - Ludwigs-Maximilian-Universität, München
- Netherlands (2):
  - Academic Ziekenhuis, Amsterdam
  - University Hospital Maastricht, Maastricht
- United Kingdom (2):
  - University of Cambridge/ Clin Med, Cambridge
  - University of Leeds, Leeds

REFERENCES:
- [Derived] Webers C, Essers I, van Tubergen A, Braun J, Heldmann F, Baraliakos X, Boonen A. Valuing Treatment With Infliximab for Ankylosing Spondylitis Using a Willingness-to-Pay Approach. Arthritis Care Res (Hoboken). 2018 Apr;70(4):608-616. doi: 10.1002/acr.23299. Epub 2018 Feb 18. PMID 28575536